CLINICAL TRIAL: NCT06337955
Title: Evolution of HCMV Non-primary Infection and Host Immune Response in HCMV-seropositive Mothers of Children Attending Day-care Centers: an Observational Prospective Study
Brief Title: Non Primary HCMV Infection: Natural History and Immune Response
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Università degli Studi di Pavia (Unknown); Merck Sharp & Dohme LLC (Industry); Fondazione Regionale per la Ricerca Biomedica (Other)
Responsible Party: Principal Investigator, Daniele Lilleri, Principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 20170007596
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, peripheral blood mononuclear cells, saliva swab, vaginal swab, urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goals of this observational study are: i) investigate the natural history of non-primary (i.e. reactivation and reinfection) HCMV infection in HCMV-seropositive Italian women and the relevant humoral and cell-mediated immune response; ii) reliably distinguish between reactivation and reinfection.

Prerequisite of the study is the availability of a maternal HCMV strain at baseline (original strain) to which subsequent strains detected during follow-up are compared in order to distinguish between reactivation (original strain) or reinfection (new strain).

To increase the likelihood of exposure to different HCMV strains, the study population is restricted to mothers of children attending day care centers.

DETAILED DESCRIPTION:
Eligible women will be identified and enrolled during pregnancy or at delivery. Consenting mothers will be tested for HCMV DNA in saliva, urine and vaginal swab at delivery and/or at the first scheduled post-partum visit (2-4 months after delivery). In addition, mothers and children will be tested for presence of HCMV DNA in milk and saliva samples, respectively.

A mother-child pair is considered HCMV-DNA positive and, therefore, suitable for continuing the study (i.e. the 12 months follow up after admission of the child to day care center) whenever viral DNA is detected in clinical samples of either the mother or the child or both. In fact, when viral DNA is undetectable in the mother but is present in the saliva of a 2-4 month old infant it can be reasonably assumed that the strain is of maternal origin.

The study does not require any modification in the normal mother-child relationship and participating mothers will be encouraged to behave normally. However, mothers will be asked to fill in a short questionnaire about basic behaviours in daily child care (i.e. frequency of hand washing, kissing of the infant, sharing of food...).

The following clinical samples will be collected from mothers and infants at indicated times (T):

T0. Delivery:

* mother: saliva, urine, vaginal swab, peripheral blood.

T1. 2-4 months after delivery:

* mother: saliva, urine, vaginal swab, milk, peripheral blood;
* infant: saliva swab.

T2. Admission of the infant to day care center:

* mother: saliva swab, urine, vaginal swab, peripheral blood;
* infant: saliva swab.

T3-T6. Every 3 months after admission of the infant for one year:

* mother: saliva swab, urine, vaginal swab, peripheral blood;
* infant: saliva swab.

Virological analyses:

1. HCMV DNA detection and quantification in blood and body specimens;
2. sequence analysis of selected variable viral genes and determination of strain(s) diversity (whole genome will also be sequenced when possible);
3. HCMV isolation from collected specimens (when HCMV DNA shedding is detected).

Immunological analyses:

* antibody response:

  1. IgG and IgM to whole HCMV antigens;
  2. IgG to glycoprotein complexes gHgLpUL128L, gHgLgO, gB;
  3. neutralizing (Nt) Ab blocking infection of epithelial/endothelial cells and fibroblasts.
* T cell response:

  1. ex vivo cytokine (IFNgamma/IL-2) production;
  2. ex vivo proliferation after stimulation with HCMV antigens;
  3. differentiation state of HCMV specific T cells (CCR7, CD45RA, IL7R expression.

Questionnaire:

Participating mothers will also be invited to fill in a questionnaire concerning their daily habits in terms of caring for their children.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) HCMV IgG-positive, breast feeding* woman.
* Willingness to enroll the infant in a public or private day care facility with at least 5 attendees at ≤ 12 months of age.
* Willingness to participate in the study.
* In case of foreign origin, language skills sufficient to understand information material and give informed consent.
* Written informed consent. * Breast feeding not required in case of availability of HCMV DNA-positive samples from the mother and/or fetus and/or newborn.

Exclusion Criteria:

* Congenital or acquired immunodeficiency
* Immunosuppressive therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be identified among pregnant women admitted for delivery at Fondazione IRCCS Policlinico San Matteo. The great majority of these women are routinely tested for HCMV antibody either in the first trimester of gestation or at the time of pre-admission for delivery at around 36 week's gestation.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HCMV non-primary infection (reinfection or reactivation). | T3-T6: 3-6-9-12 months after admission of the infant to the day-care center.
  HCMV non-primary infections will be calculated as the frequency of women with the presence of HCMV DNA in at least one of the body compartments examined (blood, saliva, urine, genital tract) at any time point. Reinfections will be considered non-primary infections in which the HCMV strain detected is different from the strain detected at baseline.

SECONDARY OUTCOMES:
HCMV-specific humoral and cell-mediated immune response during non-primary infection. | T3-T6: 3-6-9-12 months after admission of the infant to the day-care center.
  Levels of IgG and IgM to whole HCMV antigens; titers of IgG specific for HCMV envelope glycoprotein complexes; neutralizing antibody titers; number, cytokine production and proliferation of T cells in response to HCMV.
Maternal behaviours and occurrence of non-primary infection | T3-T6: 3-6-9-12 months after admission of the infant to the day-care center.
  Data collected with the questionnaire and data on HCMV shedding by the own child will be compared between women with or without non-primary infections.

OTHER OUTCOMES:
Potential use of saliva swabs for antibody determination. | T0: Enrollment.
  HCMV-specific IgG in saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Lilleri, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No